CLINICAL TRIAL: NCT00013767
Title: Child Environmental Health Center--Reducing Pesticide Exposure in Children of Farmworkers
Brief Title: Community Based Prevention/Control Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Purpose: Prevention
Other Study IDs: 9601-CP-002
Record Dates: First submitted 2001-03-29; First posted 2001-03-30 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Poisoning
Keywords: Pesticide; Insecticide; Organophosphate; Child Health; Exposure Prevention
MeSH Terms: conditions — Poisoning

INTERVENTIONS:
Behavioral: Individual and Community education

SUMMARY:
This project is aimed at better understanding how children living in agricultural environments are exposed to pesticides, and how such exposures can be prevented or reduced. The project will develop and implement a community-wide intervention to reduce the transfer of pesticides from the workplace to the home (take home pathway).

DETAILED DESCRIPTION:
This project is aimed at better understanding how children living in agricultural environments are exposed to pesticides, and how such exposures can be prevented or reduced. Since 1991 our group has investigated pesticide expsoures among children of agricultural families in Washington state, focusing on exposure to organophosphate insecticides. We have demonstrated in these studies that the residential environments of agricultural families have higher pesticide residues than do other homes in this region. We have also found that children living in these residential environments have elevated levels of pesticide metabolites in their urine. We need to better understand how these children are being exposed in order to develop recomendations for exposure prevention or reduction. The current project will develop and implement a community-wide intervention to reduce the transfer of pesticides from the workplace to the home (take home pathway). A complementary project is also underway by the UW-Child Health Center to characterize pesticide exposure pathways for children of farmworkers.

ELIGIBILITY:
Each family recruited must include one child between the ages of 1-5. Recruitment will be confined to the lower Yakima Valley.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 1999-06; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)